CLINICAL TRIAL: NCT01447017
Title: A Randomised, Parallel-group, Double-blind, Placebo-controlled Study of DPK-060 to Investigate Clinical Safety and Efficacy in Patients With Acute External Otitis
Brief Title: A Study of DPK-060 to Investigate Clinical Safety and Efficacy in Patients With Acute External Otitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DermaGen AB (Industry)
Collaborators: Pergamum AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCS-002; 2011-004356-20 (EudraCT Number)
Record Dates: First submitted 2011-09-22; First posted 2011-10-05 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-10

CONDITIONS: Acute Otitis Externa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- DPK-060 2% ear drops (Experimental): DPK-060 2% ear drops, 0.3 mL/pipette, 3 times daily for 7 or 10 days (as applicable).
  Interventions: Drug: DPK-060
- Placebo for DPK-060 ear drops (Placebo Comparator): Placebo for DPK-060 ear drops, 0.3 mL/pipette, 3 times daily for 7 or 10 days (as applicable).
  Interventions: Drug: Placebo for DPK-060 ear drops

INTERVENTIONS:
Drug: DPK-060 — DPK-060 2% ear drops were administered as 3 applications per day into the outer ear by use of a single-dose pipette (0.3 mL/pipette) for 7 days. In case clinical symptoms remained after 7 days of treatment, the treatment period was extended by another 3 days with 3 applications per day.
  Arms: DPK-060 2% ear drops
Drug: Placebo for DPK-060 ear drops — Placebo for DPK-060 ear drops were administered as 3 applications per day into the outer ear by use of a single-dose pipette (0.3 mL/pipette) for 7 days. In case clinical symptoms remained after 7 days of treatment, the treatment period was extended by another 3 days with 3 applications per day.
  Arms: Placebo for DPK-060 ear drops

SUMMARY:
The primary objective of this study is to evaluate safety and tolerability of DPK-060 2% ear drops compared to placebo for DPK-060 ear drops in patients with acute external otitis. The secondary objectives are to evaluate clinical cure and microbiological growth following treatment with DPK-060 2% ear drops compared to placebo for DPK-060 ear drops.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of acute external otitis of a severity degree not requiring specialist care
* Age 12 years and older

Exclusion Criteria:

* Known or suspected perforation of the tympanic membrane
* A clinical diagnosis of chronic suppurative otitis media, acute otitis media, acute otorrhea or malignant otitis externa
* Local ear canal abnormalities
* Congenital abnormalities of the external auditory canal or obstructive bony exostosis
* Mastoiditis or suppurative non-infectious ear disorders (e.g. cholesteatoma)
* Malignant tumour of the external auditory canal
* History of otologic surgery (except for surgery confined to the temporomandibular joint)
* Seborrheic dermatitis or other dermatological conditions of the external auditory canal that would complicate evaluation
* Current or prior use (within 7 days) of ear washes using alcohol, vinegar or other astringents
* Any clinically relevant past or present infectious/viral disease
* Current infection requiring systemic antimicrobial therapy
* Current or prior use of systemic (within 14 days) or topical (within 7 days) antibiotics
* Current or prior use of systemic (within 30 days) or topical (within 7 days) steroids
* History of immune dysfunction/deficiency and immunosuppressive therapy
* Diabetes mellitus

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Liu, MD, Principal Investigator — S3 Clinical Research Center, Vällingby; Andrzej Sloma, MD, Principal Investigator — Värmdö vårdcentral; Dan Curiac, MD, Principal Investigator — Me3+ Clinical Trials, Gothenburg; Ali Hajimirsadeghi, MD, Principal Investigator — Hagakliniken, Gothenburg; Anders Luts, MD, Principal Investigator — ProbarE, Lund; Finn Jörgensen, MD, Principal Investigator — Halmstad Lasarett ÖNH Mottagningen; Madeleine Cosmo, MD, Principal Investigator — Curakliniken, Öronmottagningen, Malmö
Locations (7):
- Sweden (7):
  - Hagakliniken, Gothenburg
  - Me3+ Clinical Trials, Gothenburg
  - Hallands Sjukhus, Halmstad
  - ProbarE, Lund
  - Curakliniken, Malmo
  - S3 Clinical Research Center, Vällingby, Stockholm
  - Värmdö vårdcentral, Stockholm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female patients, aged 12 years and above, with a clinical diagnosis of acute external otitis of a severity that is normally treated by primary care were included in the study. The first patient entered the study on January 2012 and the last patient completed the study on November 2012
Period: Overall Study
Arm/Group | DPK-060 2% Ear Drops | Placebo for DPK-060 Ear Drops
Started | 45 | 24
Performed Visit 2 | 43 | 24
Completed | 35 (In safety analysis: 42. In efficacy analyses: 40 in full analysis set, and 39 in per-protocol set.) | 14 (In safety analysis: 24. In efficacy analyses: 24 in full analysis set, and 22 in per-protocol set.)
Not Completed | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DPK-060 2% Ear Drops | Placebo for DPK-060 Ear Drops | Total
Number analyzed (Participants) | 45 | 24 | 69
Age Continuous [Mean (Standard Deviation); unit: years] — Based on the Full Analysis Set
  years | 55.0 (16.8) | 58.1 (12.3) | 56.2 (15.3)
Gender [Number; unit: participants] — Based on the Full Analysis Set
  participants
    Female | 26 | 13 | 39
    Male | 14 | 11 | 25
Region of Enrollment [Number; unit: participants]
  Sweden | 45 | 24 | 69

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (AEs)
Description: AEs were collected by a non-leading question such as "have you experienced any new health problems or worsening of existing conditions" as well as reporting events directly observed or spontaneously volunteered by patients. All AEs including but not limited to events reported by the patient, or reported in answer to an open question by the Investigator or member of the study team were recorded as an AE including the following information: Diagnosis; Start date (and time, if relevant), Stop date (and time, if relevant) or resolution; Severity; Action taken; Causality; Seriousness; Outcome.
Time Frame: AEs occurring during the treatment period were collected on day 8 or 11, as applicable. Four weeks after the last dose of investigational medicinal product (IMP), previously reported AEs were followed up and assessed as "recovered" or "not recovered".
Population: All safety analyses were performed on safety analysis set. All randomised patients who received at least 1 dose of the IMP and had at least 1 safety follow-up performed were included in the safety analysis set.
Measure: Number; unit: participants
Groups:
- DPK-060 2% Ear Drops: Patients randomized to treatment with DPK-060 2% ear drops (0.3 mL/pipette, 3 times daily for 7 or 10 days, as applicable)
- Placebo for DPK-060 Ear Drops: Patients randomized to treatment with Placebo for DPK-060 ear drops (0.3 mL/pipette, 3 times daily for 7 or 10 days, as applicable)
Arm/Group | DPK-060 2% Ear Drops | Placebo for DPK-060 Ear Drops
Number analyzed (Participants) | 42 | 24
participants
  Number patients with at least one AE | 10 | 3
  Number of patients with at least one related AE | 6 | 1
  Number patients with at least one SAE | 0 | 0
  Number of patients who withdrew due to AE | 1 | 0

ADVERSE EVENTS:
Time Frame: AEs occurring during the treatment period were collected on day 8 or 11, as applicable. Four weeks after the last dose of investigational product, previously reported AEs were followed up and assessed as "recovered" or "not recovered"
Arm/Group | DPK-060 2% Ear Drops | Placebo for DPK-060 Ear Drops
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/24
Other Adverse Events (participants affected / at risk) | 4/42 | 2/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DPK-060 2% Ear Drops (N=42) | Placebo for DPK-060 Ear Drops (N=24)
Application site pain (General disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The following disclosure restriction on the PI was included in clinical study protocol:

"If an Investigator wishes to publish results from this clinical study, written permission to publish must be obtained from the Sponsor in advance. As some of the information regarding the IP and development activities at the Sponsor may be of a strictly confidential nature, the Sponsor must first review any publication manuscript prior to their submission to journals, meetings or conferences."